CLINICAL TRIAL: NCT06859060
Title: Testing Bridges to Better Health and Wellness for People Living With Serious Mental Illness in Puerto Rico
Brief Title: Improving Health and Wellness for People With Serious Mental Illness in Puerto Rico
Acronym: BRIDGES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ponce Medical School Foundation, Inc. (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2308159485; 2U54MD007579-39 (NIH)
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Chronic Disease; Serious Mental Illness
Keywords: Bridges; Stigma; Preventive Primary Care; Healthcare Managers; Wellness
MeSH Terms: conditions — Chronic Disease; Social Stigma

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BRIDGES Intervention (Experimental): Participants randomized to the experimental condition will receive the BRIDGES Healthcare Manager Intervention.
  Interventions: Behavioral: BRIDGES Healthcare Manager Intervention
- Enhanced Treatment as Usual (ETAU) (Other): Participants randomized to the control condition will receive standard psychiatric care with an informational brochure on accessing primary care providers.
  Interventions: Other: Enhanced Treatment as Usual (ETAU)

INTERVENTIONS:
Behavioral: BRIDGES Healthcare Manager Intervention — A culturally adapted, multilevel intervention consisting of monthly 60-minute sessions over a 12-month period. Sessions will be conducted by graduate clinical psychology students acting as healthcare managers. The intervention focuses on care coordination, patient activation, and reducing provider stigma to improve access to preventive primary care services.
  Arms: BRIDGES Intervention
Other: Enhanced Treatment as Usual (ETAU) — Participants will continue to receive standard psychiatric care, including routine visits with their mental health providers at the designated clinical sites. They will also receive a booklet with information on how best to link with primary care providers. This ensures that participants are aware of available resources and basic health care recommendations, but does not include any active follow-up or intervention components.
  Arms: Enhanced Treatment as Usual (ETAU)

SUMMARY:
This study evaluates the effectiveness of a culturally tailored intervention, Bridges to Better Health and Wellness (BRIDGES), aimed at reducing chronic disease disparities among Puerto Ricans with serious mental illness (SMI). Participants receive monthly sessions with health care managers to address patient-provider stigma and care coordination.

DETAILED DESCRIPTION:
BRIDGES is a multi-level Healthcare Manager Intervention (HMI) that addresses both patient and provider barriers to healthcare. It includes culturally adapted modules to reduce stigma and promote chronic disease prevention. The study uses a hybrid type 1 effectiveness-implementation randomised controlled trial to test its impact on primary care service use, chronic disease outcomes and stigma reduction over 12 months.

ELIGIBILITY:
Inclusion criteria:

Adults receiving psychiatric or psychological services at the Wellness Center or the Mayaguez Medical Center - Primary Care Diagnosed with at least one serious mental illness SMI (e.g., schizophrenia, bipolar disorder, major depression, etc.) Have at least one risk factor or a diagnosis of a chronic health condition (e.g., diabetes, overweight, hypertension, etc.).

Be willing to receive or continue preventive medical care with a primary care physician.

Exclusion criteria:

Have started psychiatric or mental health services at least one month before Have been diagnosed with a general mental health condition (e.g., Depression or Anxiety).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Recipt of Preventive Primary Care | baseline,6 and 12 months follow up and 6 and 12 months post intervention
  29-item questionnaire developed by team members. It uses preventive primary care indicators from the US Preventive Service Task Force Guidelines extracted from medical records and examines the use of physical health services over the past 6-months.Indicators are grouped into six categories: physical examinations, screenings for women, screenings for men, laboratory tests, vaccinations, and education. An aggregate preventive primary score is calculated representing the proportion of services for which each participant was eligible depending on age and gender.

SECONDARY OUTCOMES:
Hemoglobin A1c | baseline,6 and 12 months follow up and 6 and 12 months post intervention
  The A1C test is a simple common blood test used to measure blood sugar levels over the past 3 months.
Lipid Panel | baseline,6 and 12 months follow up and 6 and 12 months post intervention
  The Lipid panel is a simple common blood test used to examine cardiovascular health by analyzing cholesterol in the blood. This test examines four types of lipids in the blood, namely: 1) Total cholesterol, 2 Low-density lipoprotein (LDL), 3) High-density lipoprotein (HDL), and 4) Triglycerides.
Basic Metabolic Panel | baseline,6 and 12 months follow up and 6 and 12 months post intervention
  It is a simple common blood group of tests used to examine different naturally occurring chemicals in the blood. The tests can give information heart, kidneys, and liver function. It includes Blood urine nitrogen (BUN), carbon dioxide (C02), Creatinine, Glucose, Serum chloride, Serum potassium, Serum sodium, and Serum Calcium.
Smoking - Severity Dependence Scale | baseline,6 and 12 months follow up and 6 and 12 months post intervention
  Five-item scale, used to assess severity of smoking.
Physical Activity - International Physical Activity Questionnaire | baseline,6 and 12 months follow up and 6 and 12 months post intervention
  This is a 7-item measure widely used to examine 4 types of physical activity: 1) vigorous, 2) moderate, 3) walking and 4) sitting.
Health Literacy - Test of Functional Health Literacy for Adults | baseline,6 and 12 months follow up and 6 and 12 months post intervention
  Questionnaire with 12 items measuring adult functional health literacy in the health care setting.
Self-Stigma - Self-Stigma of Mental Illness Scale | baseline,6 and 12 months follow up and 6 and 12 months post intervention
  This 40-item measure examines self stigma's four dimensions (awareness, agreement, self-application and self esteem).
Provider Stigma - The Mental Health Stigma Scale for Health Professionals | baseline,6 and 12 months follow up and 6 and 12 months post intervention
  12-item measure examining provider stigma dimensions (social distance, negative character attributions and self-sufficiency).
Patient-Provider Relationship - Patient Assessment of Chronic Illness Care | baseline,6 and 12 months follow up and 6 and 12 months post intervention
  20-item scale used to assess participants' perspectives on the quality and patient-centeredness of chronic illness care received during the past 6 months from their primary care provider.

CONTACTS AND LOCATIONS:
Locations (2):
- Puerto Rico (2):
  - Mayagüez Medical Center Primary Care Psychology Clinic, Mayagüez, Puerto Rico
  - PHSU Wellness Center, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided